CLINICAL TRIAL: NCT03765931
Title: Comparative Efficacy of Single-dose Doxycycline Versus Standard 5- Day Amoxicillin Treatment for Patients With Non-malarial Fever: a Randomized Non-inferiority Trial in Senegal
Brief Title: Comparative Efficacy of Single-dose Doxycycline Versus Standard 5- Day Amoxicillin Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Principal Investigator, Aldiouma Diallo, MD, Institut de Recherche pour le Developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCTDOXY2016
Record Dates: First submitted 2018-06-20; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Doxycycline; Amoxicillin

STUDY DESIGN:
Intervention Model Description: We aimed to determine the efficacy of a single dose of doxycycline compared to a 5-day amoxicillin course for the treatment of fever.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subjects treated with doxycycline (Active Comparator): The participants treated by doxycycline 100 mg will have one dose but followed 5 days
  Interventions: Drug: Doxycycline
- subjects treated with amoxycilline (Placebo Comparator): The participants treated with amoxycilline 500 mg will have 2 doses per days during 5 days treatement and follwed during these 5 days
  Interventions: Drug: Doxycycline; Drug: Amoxicillin

INTERVENTIONS:
Drug: Doxycycline — The investigators conducted a non-inferiority, open-label, randomized controlled trial in patients aged > 8 years recruited from dispensaries in the rural area of Niakhar, Senegal. Participants were enrolled based on a body temperature > 37.5°C, as assessed using an electronic axillary thermometer. Febrile patients with a positive malaria test were excluded from the study. Participants were randomly assigned (2:1) to receive either a single dose of doxycycline (30 mg/kg) or a five-day course of amoxicillin (20 mg/kg) by a computer-generated random number sequence. The investigators monitored participants at days 2 and 7 post-treatment. The primary outcome was cure after 7 days, defined as a body temperature < 37.5°C.
Drug: Amoxicillin — The investigators conducted a non-inferiority, open-label, randomized controlled trial in patients aged > 8 years recruited from dispensaries in the rural area of Niakhar, Senegal. Participants were enrolled based on a body temperature > 37.5°C, as assessed using an electronic axillary thermometer. Febrile patients with a positive malaria test were excluded from the study. Participants were randomly assigned (2:1) to receive either a single dose of doxycycline (30 mg/kg) or a five-day course of amoxicillin (20 mg/kg) by a computer-generated random number sequence. The investigators monitored participants at days 2 and 7 post-treatment. The primary outcome was cure after 7 days, defined as a body temperature < 37.5°C.
  Arms: subjects treated with amoxycilline

SUMMARY:
Abstract: Background The current practice in Senegal is to use broad-spectrum antibiotics including amoxicillin and/or cotrimoxazole in case of non-malarial fevers. First-line treatment with doxycycline has cured such patients. The investgators aimed to determine the efficacy of a single dose of doxycycline compared to a 5-day amoxicillin course for the treatment of fever.

DETAILED DESCRIPTION:
Methods The investgators conducted a non-inferiority, open-label, randomized controlled trial in patients aged > 8 years recruited from dispensaries in the rural area of Niakhar, Senegal. Participants were enrolled based on a body temperature > 37.5°C, as assessed using an electronic axillary thermometer. Febrile patients with a positive malaria test were excluded from the study. Participants were randomly assigned (1:1) to receive either a single dose of doxycycline (30 mg/kg) or a five-day course of amoxicillin (20 mg/kg) by a computer-generated random number sequence. The investgators monitored participants at days 2 and 7 post-treatment. The primary outcome was cure after 7 days, defined as a body temperature < 37.5°C. The investgators used a non-inferiority margin of 10%. This trial was approved by the national ethic committees of the Senegalese Ministry of Health in May 2017 (0026/MSAS/DPRS/CNERS, March, 7, 2016).

ELIGIBILITY:
Inclusion Criteria:

* Participants over 8 years with no malaria fever

Exclusion Criteria:

Under 8 years Pregnanants women

-

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-07; Primary Completion 2017-01 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Non-inferiority comparison of the efficacy between Doxycycline and Amoxicillin after 7 days of follow-up | 7 days follow up
  The endpoint was cure at day-7 post-inclusion. Clinical cure was defined as a body temperature < 37.5°C. Clinical failure was defined as persistence of fever > 37.5°C at day-7. The investgators used a non-inferiority margin of 10%.

CONTACTS AND LOCATIONS:
Locations (1):
- Niakhar observational site, Niakhar, Fatick, Senegal

IPD SHARING:
Plan to Share IPD: Yes
Will share by restitution with the communuty
Supporting Information: Study Protocol, CSR
Time Frame: Just after close out and analysing the data
Access Criteria: Share with participants but also with the ministry of heath